CLINICAL TRIAL: NCT02645019
Title: The Effect of EGD Probe Insertion on the Intracuff Pressure of the Laryngeal Mask Airway or Cuffed Endotracheal Tube in Children
Status: Completed | Type: Observational
Sponsor: Mineto Kamata (Other)
Responsible Party: Sponsor-Investigator, Mineto Kamata, Anesthesia Clinical Fellow, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB15-01074
Record Dates: First submitted 2015-12-30; First posted 2016-01-01 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Esophagogastroduodensocopy (EGD) Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Cuffed ETT: Airway secured using a cuffed endotracheal tube.
  Interventions: Device: Cuffed ETT
- LMA 2: Airway secured using a size 2 laryngeal mask airway.
  Interventions: Device: Cuffed LMA
- LMA 2.5: Airway secured using a size 2.5 laryngeal mask airway.
  Interventions: Device: Cuffed LMA
- LMA 3: Airway secured using a size 3 laryngeal mask airway.
  Interventions: Device: Cuffed LMA
- LMA 4: Airway secured using a size 4 laryngeal mask airway.
  Interventions: Device: Cuffed LMA

INTERVENTIONS:
Device: Cuffed ETT — Cuffed endotracheal tube.
  Groups: Cuffed ETT
Device: Cuffed LMA — Cuffed laryngeal mask airway.
  Groups: LMA 2; LMA 2.5; LMA 3; LMA 4

SUMMARY:
A prospective study designed to access changes in the intracuff pressure of a laryngeal mask airway (LMA) or cuffed endotracheal tube (cETT) during placement of an esophagogastroduodenoscopy (EGD) probe during an EGD in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 0-18 years old having EGD procedure with a LMA or cuffed ETT.

Exclusion Criteria:

* Patients with a history of tracheomalacia, bronchomalacia or any other airway issues.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from 0-18 years old having EGD procedure with LMA or cuffed ETT.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cuffed ETT | LMA 2 | LMA 2.5 | LMA 3 | LMA 4
Started | 13 | 15 | 15 | 33 | 24
Completed | 13 | 15 | 15 | 33 | 24
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LMA 2 | LMA 2.5 | LMA 3 | LMA 4 | Cuffed ETT | Total
Number analyzed (Participants) | 15 | 15 | 33 | 24 | 13 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 33 | 24 | 13 | 100
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 19 | 10 | 7 | 52
  Male | 6 | 8 | 14 | 14 | 6 | 48
Intracuff pressure immediately following intubation [Mean (Standard Deviation); unit: cmH2O] — Population: Number of participants analyzed in each row is number that received each type of airway.
  cmH2O | 15 (13) | 25 (10) | 34 (10) | 32 (10) | 19 (26) | 27 (15)

OUTCOME MEASURES:

1. Primary Outcome: Intracuff Pressures During Probe Insertion
Description: Intracuff pressure in cmH2O of cuffed ETT or LMA during EGD probe insertion.
Time Frame: At time of EGD probe insertion
Population: Number of participants that received each type of airway.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | LMA 2 | LMA 2.5 | LMA 3 | LMA 4 | Cuffed ETT
Number analyzed (Participants) | 15 | 15 | 33 | 24 | 13
cmH2O | 22 (14) | 34 (9) | 41 (15) | 37 (12) | 24 (25)

2. Primary Outcome: Intracuff Pressure With Probe in Place
Description: Intracuff pressure in cmH2O of cuffed ETT or LMA during EGD while probe is in place.
Time Frame: At time of EGD while probe is in place
Population: Number of participants analyzed in each row is number that received each type of airway.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | LMA 2 | LMA 2.5 | LMA 3 | LMA 4 | Cuffed ETT
Number analyzed (Participants) | 15 | 15 | 33 | 24 | 13
cmH2O | 22 (14) | 35 (9) | 39 (13) | 36 (11) | 24 (25)

3. Primary Outcome: Intracuff Pressure After Probe Removal
Description: Intracuff pressure in cmH2O of cuffed ETT or LMA after EGD probe is removed.
Time Frame: Immediately after probe removal
Population: Number of participants analyzed in each row is number that received each type of airway.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | LMA 2 | LMA 2.5 | LMA 3 | LMA 4 | Cuffed ETT
Number analyzed (Participants) | 15 | 15 | 33 | 24 | 13
cmH2O | 15 (11) | 26 (10) | 31 (11) | 29 (10) | 21 (25)

ADVERSE EVENTS:
Arm/Group | LMA 2 | LMA 2.5 | LMA 3 | LMA 4 | Cuffed ETT
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/33 | 0/24 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/33 | 0/24 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/33 | 0/24 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes